CLINICAL TRIAL: NCT01173315
Title: The Impact of Vitamins and Minerals Supplementation on Neuropathy and Nephropathy Complications in Type 2 Diabetic Patients: a Randomised Clinical Trial
Brief Title: The Impact of Vitamins and Minerals Supplementation on Neuropathy and Nephropathy Complications
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Dr Majid Hajifaraji, National Nutrition and Food Technology Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MFarvid
Record Dates: First submitted 2010-07-30; First posted 2010-08-02 (Estimated); Last update posted 2010-08-02 (Estimated); Status verified 2006-04

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; micronutrients; nephropathy; neuropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Kidney Diseases | interventions — Vitamins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Group MV (Experimental): Group MV: Zinc sulfate and Magnesium oxide (providing 10 mg Zn and 125 mg Mg) and vitamin C (100 mg) and vitamin E (100 mg
  Interventions: Dietary Supplement: vitamin and mineral supplementation
- Group MVB (Experimental): Group MVB: Zinc sulfate and Magnesium oxide (providing 10 mg Zn and 125 mg Mg) and vitamin C (100 mg) and vitamin E (100 mg)plus vitamin B1 (5 mg), vitamin B2 (5 mg), vitamin B6 (5 mg), biotin (50 µg), vitamin B12 (5 µg) and folic acid (0.5 mg)
  Interventions: Dietary Supplement: vitamin and mineral supplementation
- Group P (Placebo Comparator): Group P: starch (placebo
  Interventions: Dietary Supplement: vitamin and mineral supplementation

INTERVENTIONS:
Dietary Supplement: vitamin and mineral supplementation — Group MV: Zinc sulfate and Magnesium oxide (providing 10 mg Zn and 125 mg Mg) and vitamin C (100 mg) and vitamin E (100 mg); Group MVB: both of the above mineral and vitamin supplements plus vitamin B1 (5 mg), vitamin B2 (5 mg), vitamin B6 (5 mg), biotin (50 µg), vitamin B12 (5 µg) and folic acid (0.5 mg); Group P: starch (placebo).

SUMMARY:
The combination of vitamin and mineral supplementation may improve:

* glycemic control
* lipid profile
* oxidative stress
* blood pressure
* nephropathy indices
* neuropathy indices

DETAILED DESCRIPTION:
A total of 75 diabetic patients (39 men and 36 women), aged 36 to 69 years, having diabetes for at least 3 years, was recruited for this study. Type 2 diabetes was defined as fasting plasma glucose 126 mg/dl (two times repeated) or taking oral glucose-lowering agents.Diabetic patients were stratified by sex and randomly assigned to one of the three treatment groups using block randomization procedure. Depending upon the treatment groups, each subject received two capsules per day, 1 with breakfast and 1 with dinner, for a period of 4 months. Each capsule contained one of the following preparations and hence determined the corresponding groups: Group MV: Zinc sulfate and Magnesium oxide (providing 10 mg Zn and 125 mg Mg) and vitamin C (100 mg) and vitamin E (100 mg); Group MVB: both of the above mineral and vitamin supplements plus vitamin B1 (5 mg), vitamin B2 (5 mg), vitamin B6 (5 mg), biotin (50 µg), vitamin B12 (5 µg) and folic acid (0.5 mg); Group P: starch (placebo). All of the study medications, including the placebo, were supplied by Pharmaceutical Sciences Research Center (Tehran University of Medical Sciences, Iran) and were indistinguishable from each other. They were stored at 20-25 0C.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for 3 years

Exclusion Criteria:

* Resting blood pressure >160/100 mmHg
* Taking vitamin and/or mineral supplement, thyroid hormones, estrogens, progesterone, diuretics or antihypertensive agents
* Having history of myocardial infarction and hepatic disease
* Pregnant

Ages: 30 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-06; Primary Completion 2008-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Evidence of clinically neuropathy confirmed by nerve conduction velocities | 4 months
  nerve conduction velocities in the bilateral sural sensory nerves, and peroneal, tibial, median, and ulnar motor nerves with F waves in hands and legs extremity

SECONDARY OUTCOMES:
nephropathy indices were determined by 3 times urine microalbumin concentration using Enzyme Immuno Assay commercial kit | 4 months
  Urine microalbumin concentration was measured by Enzyme Immuno Assay using commercial kit (ORG 5MA Micro Albumin, Orgentec Diagnostika GmbH, and Mainz, Germany). Urine total protein was determined by lowry method (19). Urine samples creatinine (Cr) were measured by chemical colorimetric kit according Jaffe reaction (Pars Azmoun, Tehran, Iran) and all urine results were expressed in relation to gram creatinine excretion.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Sadat Farvid, Ph.D., Principal Investigator — Shahid Beheshti University of Medical Sciences

REFERENCES:
- [Derived] Farvid MS, Homayouni F, Amiri Z, Adelmanesh F. Improving neuropathy scores in type 2 diabetic patients using micronutrients supplementation. Diabetes Res Clin Pract. 2011 Jul;93(1):86-94. doi: 10.1016/j.diabres.2011.03.016. Epub 2011 Apr 14. PMID 21496936